CLINICAL TRIAL: NCT04985552
Title: Closed Incision Negative Pressure Therapy Compared to Conventional Dressing Following Autologous Abdominal Tissue Breast Reconstruction: A Pilot Randomized Control Trial
Brief Title: ciNPT in Autologous Abdominal Tissue Breast Reconstruction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13155
Record Dates: First submitted 2021-07-05; First posted 2021-08-02 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- ciNPT (Experimental)
  Interventions: Procedure: DIEP Breast Reconstruction; Device: ciNPT
- Conventional tape dressings (Active Comparator)
  Interventions: Procedure: DIEP Breast Reconstruction; Other: Conventional Tape Dressings

INTERVENTIONS:
Procedure: DIEP Breast Reconstruction — All patients enrolled in the study will undergo DIEP breast reconstruction and have their abdominal incision sutured according to routine clinical practice: 3-0 VICRYL ® suture (Ethicon, USA) for deep fascia closure, 4-0 MONOCRYL® suture (Ethicon, USA) for deep dermal closure, and 5-0 MONOCRYL® suture (Ethicon, USA) for subcuticular closure.
Device: ciNPT — Following closure of the abdominal donor site, the closed incision will be dressed with the ciNPT system [V.A.C.ULTA™ Negative Pressure Wound Therapy System (KCI, USA)] applied by the operating surgeon in a sterile fashion. The ciNPT device will be set at -125mmHg of continuous negative pressure for a period of 7 days or until patient discharge from hospital. Removal of the ciNPT dressing will be performed by the surgical team at the time of discharge. Following removal, no additional dressings will be applied to the abdominal incision unless clinically indicated secondary to dehiscence.
  Arms: ciNPT
Other: Conventional Tape Dressings — Following closure of the abdominal donor site, the closed abdominal incision will be dressed with 1-inch Micropore™ Surgical Tape (3M, USA) with an alcohol swab applied to the tape for additional adhesion, by the operating surgeon in a sterile fashion. This dressing will remain in-situ for up to 7 days or until patient discharge from hospital. Removal of the traditional tape dressing will be performed by the surgical team at the time of discharge. Following removal, no additional dressings will be applied unless clinically indicated secondary to dehiscence.
  Arms: Conventional tape dressings

SUMMARY:
In women who undergo mastectomy for the treatment of breast cancer, autologous reconstruction using the deep inferior epigastric perforator (DIEP) flap is a common surgical procedure that aims to restore both the appearance and texture of the breast(s). Specifically, this requires the transfer of skin, fat, and perforator vessels from the abdomen to a recipient artery and vein in the chest to create a viable breast mound. Post-operatively, the abdominal donor site is routinely monitored for wound dehiscence, which has a reported incidence of up to 39% in this patient population; however, this incidence typically varies from 3.5% to 14%.

At the investigators' academic institution, patients who undergo DIEP breast reconstruction typically have closed incision negative pressure therapy (ciNPT) or traditional tape dressings applied to the closed abdominal donor site. These dressings are selected according to surgeon preference and typically remain in-situ until hospital discharge. As there remains clinical equipoise regarding the ability of ciNPT to reduce abdominal wound dehiscence, further research in the form of a parallel, two-arm RCT is warranted.

The investigators propose a pilot study comparing ciNPT to standard tape dressings to the abdominal donor site incision for patients undergoing autologous DIEP breast reconstruction. As a pilot trial, the primary objective of the study is to assess feasibility outcomes. The design and conduct of the proposed pilot study will mirror the methodology of the definitive trial including randomization, interventions, and clinical outcomes. The secondary objective of this study is to evaluate clinical outcomes comparing ciNPT to standard tape dressings applied to the abdominal donor site incision. Clinical outcomes will include: 1) the incidence of abdominal wound dehiscence at 4 weeks following DIEP breast reconstruction; 2) the incidence of seroma formation and surgical site infection at 4 weeks; 3) quality of life as measured by BREAST-Q physical well-being abdomen and EQ-5D-5L pre-operatively, 1-month, 6-months, and 12-months postoperatively; 4) Scar appearance as measured by the SCAR-Q at 12-months postoperatively.

The pilot RCT will demonstrate feasibility of a definitive trial comparing ciNPT to standard tape dressings for the abdominal donor site of patients undergoing DIEP breast reconstruction. A priori hypotheses for each feasibility outcome will be:

1. Eligibility: At least 90% of screened patients will be eligible.
2. Recruitment: At least 85% of eligible patients will be enrolled. To be considered fully enrolled patients must sign the informed consent form, complete baseline demographic questionnaires, and be randomized to a study arm.
3. Retention: At least 85% of randomized patients will complete the study, defined as completion of 12-month follow-up

ELIGIBILITY:
Inclusion Criteria:

* adult female patients (≥ 18 years old)
* consent to elective immediate (i.e. performed at the time of mastectomy) or delayed (i.e. performed following mastectomy) breast reconstruction using the DIEP flap

Exclusion Criteria:

* patients who are pregnant
* have a documented/reported allergy to adhesive dressings

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of Patient Eligibility - Study Feasibility | 12 months
  The percentage of patients that are eligible for the study among those that are screened will be recorded. This criteria will be determined to be feasible if at least 90% of screened patients are deemed to be eligible.
Percentage of Patient Recruitment - Study Feasibility | 12 months
  The percentage of patients that are enrolled in the study among those determined to be eligible will be recorded. To be considered fully enrolled patients must sign the informed consent form, complete baseline demographic questionnaires, and be randomized to a study arm. This criteria will be determined to be feasible if at least 85% of eligible patients are recruited.
Percentage of Patient Retention - Study Feasibility | 12 months
  The percentage of patients that complete the study among those that are randomized will be recorded. Completion of the study will be defined as completion of 12 month follow-up questionnaires. This criteria will be determined to be feasible if at least 85% of randomized patients complete the study.
  As per Thabane et al., the investigators will collate the results of all three of the aforementioned primary outcomes to determine study eligibility. If all three criteria are met, the authors will decide that the study is feasible and continue without modifications. If one or more criteria is not met, the investigators will either decide to:
  Stop - main study not feasible, or Continue, but modify protocol - feasible with modifications, or Continue without modifications, but monitor closely - feasible with close monitoring

SECONDARY OUTCOMES:
Percentage of participants with Abdominal Wall Dehiscence | 4 weeks
  the between-group difference in the incidence of abdominal wound dehiscence- 'wound dehiscence' will be defined as the partial or full-thickness separation of the abdominal wound incision necessitating routine dressing changes, surgical debridement, or revision of the abdominal incision
Percentage of participants with Seroma Formation | 4 weeks
  seroma formation - defined by the presence of a symptomatic, subcutaneous fluid collection (diagnosed clinically or by ultrasound per clinician judgement)
Percentage of participants with Surgical Site Infection | 4 weeks
  surgical site infection - necessitating antibiotic administration (diagnosed clinically or by wound swab)
5-level EQ-5D version (EQ-5D-5L) - Patient Quality of Life | 12 months
  The EQ-5D-5L essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). This scale is a patient-reported outcome measure (PROM) designed to measure overall health status. The EQ-5D measures 5 health states measured from 1-5, with 1 being the best and 5 being the worst. An overall score can be generated from this with the best health at the minimum score of 5, and the worst health state at the maximum score of 25. The EQ VAS is an analogue scale from 0-100, with 100 being the best health and 0 being the worst health that you can imagine.
BREAST-Q physical well-being abdomen - Patient Quality of Life | 12 months
  The BREAST-Q physical well-being abdomen is a patient-reported outcome measure (PROM) designed to measure the negative physical sequelae of the abdomen following autologous tissue reconstruction. Total scores are converted to an equivalent Rasch transformed score from 0 to 100. 0 represents the worst outcome and 100 represents the best outcome.
SCAR-Q - Patient Quality of Life | 12 months
  The BREAST-Q physical well-being abdomen is a patient-reported outcome measure (PROM) designed to measure the the appearance, symptoms, and psychosocial impact of scars. Total scores are converted to an equivalent Rasch transformed score from 0 to 100. 0 represents the worst outcome and 100 represents the best outcome.

REFERENCES:
- [Background] Leyngold MM. Is Unipedicled Transverse Rectus Abdominis Myocutaneous Flap Obsolete Owing to Superiority of DIEP Flap? Ann Plast Surg. 2018 Jun;80(6S Suppl 6):S418-S420. doi: 10.1097/SAP.0000000000001319. PMID 29369109
- [Background] Chang EI, Liu J. Prospective Evaluation of Obese Patients Undergoing Autologous Abdominal Free Flap Breast Reconstruction. Plast Reconstr Surg. 2018 Aug;142(2):120e-125e. doi: 10.1097/PRS.0000000000004550. PMID 29794640
- [Background] Muller-Sloof E, de Laat HEW, Hummelink SLM, Peters JWB, Ulrich DJO. The effect of postoperative closed incision negative pressure therapy on the incidence of donor site wound dehiscence in breast reconstruction patients: DEhiscence PREvention Study (DEPRES), pilot randomized controlled trial. J Tissue Viability. 2018 Nov;27(4):262-266. doi: 10.1016/j.jtv.2018.08.005. Epub 2018 Aug 14. PMID 30126630
- [Background] Lindenblatt N, Gruenherz L, Farhadi J. A systematic review of donor site aesthetic and complications after deep inferior epigastric perforator flap breast reconstruction. Gland Surg. 2019 Aug;8(4):389-398. doi: 10.21037/gs.2019.06.05. PMID 31538064
- [Background] Thacoor A, Kanapathy M, Torres-Grau J, Chana J. Deep inferior epigastric perforator (DIEP) flap: Impact of drain free donor abdominal site on long term patient outcomes and duration of inpatient stay. J Plast Reconstr Aesthet Surg. 2018 Aug;71(8):1103-1107. doi: 10.1016/j.bjps.2018.04.019. Epub 2018 May 22. PMID 29910106
- [Background] Nelson JA, Chung CU, Fischer JP, Kanchwala SK, Serletti JM, Wu LC. Wound healing complications after autologous breast reconstruction: a model to predict risk. J Plast Reconstr Aesthet Surg. 2015 Apr;68(4):531-9. doi: 10.1016/j.bjps.2014.11.017. Epub 2014 Nov 28. PMID 25557724
- [Background] Sandy-Hodgetts K, Watts R. Effectiveness of negative pressure wound therapy/closed incision management in the prevention of post-surgical wound complications: a systematic review and meta-analysis. JBI Database System Rev Implement Rep. 2015 Jan;13(1):253-303. doi: 10.11124/jbisrir-2015-1687. PMID 26447018
- [Background] Wilkes RP, Kilpad DV, Zhao Y, Kazala R, McNulty A. Closed incision management with negative pressure wound therapy (CIM): biomechanics. Surg Innov. 2012 Mar;19(1):67-75. doi: 10.1177/1553350611414920. Epub 2011 Aug 25. PMID 21868417
- [Background] Hyldig N, Birke-Sorensen H, Kruse M, Vinter C, Joergensen JS, Sorensen JA, Mogensen O, Lamont RF, Bille C. Meta-analysis of negative-pressure wound therapy for closed surgical incisions. Br J Surg. 2016 Apr;103(5):477-86. doi: 10.1002/bjs.10084. PMID 26994715
- [Background] Tran BNN, Johnson AR, Shen C, Lee BT, Lee ES. Closed-Incision Negative-Pressure Therapy Efficacy in Abdominal Wall Reconstruction in High-Risk Patients: A Meta-analysis. J Surg Res. 2019 Sep;241:63-71. doi: 10.1016/j.jss.2019.03.033. Epub 2019 Apr 19. PMID 31009887
- [Background] Siegwart LC, Sieber L, Fischer S, Maraka S, Kneser U, Kotsougiani-Fischer D. Influence of closed incision negative-pressure therapy on abdominal donor-site morbidity in microsurgical breast reconstruction. Microsurgery. 2022 Jan;42(1):32-39. doi: 10.1002/micr.30683. Epub 2020 Nov 17. PMID 33201541
- [Background] Little RJ, D'Agostino R, Cohen ML, Dickersin K, Emerson SS, Farrar JT, Frangakis C, Hogan JW, Molenberghs G, Murphy SA, Neaton JD, Rotnitzky A, Scharfstein D, Shih WJ, Siegel JP, Stern H. The prevention and treatment of missing data in clinical trials. N Engl J Med. 2012 Oct 4;367(14):1355-60. doi: 10.1056/NEJMsr1203730. No abstract available. PMID 23034025
- [Background] Whitehead AL, Julious SA, Cooper CL, Campbell MJ. Estimating the sample size for a pilot randomised trial to minimise the overall trial sample size for the external pilot and main trial for a continuous outcome variable. Stat Methods Med Res. 2016 Jun;25(3):1057-73. doi: 10.1177/0962280215588241. Epub 2015 Jun 19. PMID 26092476
- [Background] Eldridge SM, Lancaster GA, Campbell MJ, Thabane L, Hopewell S, Coleman CL, Bond CM. Defining Feasibility and Pilot Studies in Preparation for Randomised Controlled Trials: Development of a Conceptual Framework. PLoS One. 2016 Mar 15;11(3):e0150205. doi: 10.1371/journal.pone.0150205. eCollection 2016. PMID 26978655
- [Background] Thoma A, Avram R, Dal Cin A, Murphy J, Duku E, Xie F. Cost-effectiveness Analysis of Abdominal-based Autogenous Tissue and Tissue-expander Implant following Mastectomy. Plast Reconstr Surg Glob Open. 2020 Apr 11;8(10):e2986. doi: 10.1097/GOX.0000000000002986. eCollection 2020 Oct. PMID 33173657
- [Background] Thoma A, Avram R, Dal Cin A, Murphy J, Duku E, Xie F. Comparing the Clinical and Cost-Effectiveness of Abdominal-based Autogenous Tissue and Tissue-Expander Implant: A Feasibility Study. Plast Reconstr Surg Glob Open. 2020 Apr 11;8(10):e3179. doi: 10.1097/GOX.0000000000003179. eCollection 2020 Oct. PMID 33173691
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Derived] Gallo L, Kim P, Dunn E, Churchill I, Yuan M, Avram R, McRae M, Thoma A, Coroneos CJ, Voineskos SH. Closed-Incision Negative Pressure Therapy Compared to Conventional Dressing Following Autologous Abdominal Tissue Breast Reconstruction: The MACVAC Pilot Randomized Control Trial. Plast Surg (Oakv). 2025 Jul 1:22925503251350926. doi: 10.1177/22925503251350926. Online ahead of print. PMID 40611914
- See also: The World Union of Wound Healing Societies (WUWHS) defines surgical wound dehiscence as "all degrees of separation of the margins of a closed surgical incision". — https://www.woundsinternational.com/resources/details/consensus-document-surgical-wound-dehiscence-improving-prevention-and-outcomes
- See also: Related Info — https://www.ema.europa.eu/en/documents/scientific-guideline/guideline-missing-data-confirmatory-clinical-trials_en.pdf
- See also: EQ-5D-5L — https://euroqol.org/publications/user-guides
- See also: BREAST-Q — http://qportfolio.org/wp-content/uploads/2020/02/BREAST-Q-USERS-GUIDE-V2.pdf
- See also: SCAR-Q — http://qportfolio.org/wp-content/uploads/2020/02/SCAR-Q-USERS-GUIDE-V1.pdf